CLINICAL TRIAL: NCT00144404
Title: Baseline Sexual Function, Cognitive Function, Body Composition and Muscle Parameters and Pharmacokinetics of Transdermal Testosterone Gel in Women With Hypopituitarism
Status: Withdrawn | Type: Observational
Why Stopped: this was not a clinical trial
Sponsor: Charles Drew University of Medicine and Science (Other)
Responsible Party: Theodore C. Friedman, M.D., Ph.D. Principal Investigator, Charles Drew University of Medicine and Science
Other Study IDs: 02-04-376-07
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Panhypopituitarism
MeSH Terms: conditions — Combined Pituitary Hormone Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine the blood levels of testosterone gel administered for a week to women with hypopituitarism and determine if this leads to testosterone replacement in a normal range for women. An additional objective is to determine the baseline laboratory abnormalities and physical, brain function, emotional and sexual symptomatology of these women with hypopituitarism.

DETAILED DESCRIPTION:
The ovaries and the adrenal glands contribute to the daily production of 300 micrograms of testosterone in healthy, menstruating women. The physiologic role of testosterone in women, however, remains poorly understood. Previous studies of testosterone supplementation, largely in surgically or naturally menopausal women, have reported improvements in subjective measures of sexual function, sense of well being, and variable changes in markers of bone formation and resorption. However, many of these previous studies used supraphysiologic doses of testosterone, and insensitive assays for the measurement of total and free testosterone levels that lacked precision and accuracy in the low range prevalent in women. The effects of testosterone in women on body composition, muscle performance and physical function have not been studied. Therefore, the clinical significance of androgen deficiency in women remains unclear. Thus, we do not know whether physiologic testosterone replacement of women with androgen deficiency can produce clinically meaningful improvements in sexual and cognitive functions, fat-free mass, and muscle performance, without virilizing side effects.

Women with hypopituitarism represent an excellent model to study the effects of physiologic replacement as these patients have severely diminished androgen production from both the adrenal glands and the ovaries. Estrogen administration, by increasing sex hormone binding globulin (SHBG) in these women leads to further reduction in free testosterone concentrations. In fact, a recent study demonstrated very low levels of total and free testosterone, dehydroepiandrosterone sulfate (DHEAS), its parent steroid dehydroepiandrosterone (DHEA), and androstenedione in women with hypopituitarism. Therefore, it is postulated that many women with hypopituitarism suffer from decreased libido, altered body composition, and impaired quality of life, symptoms possibly related to androgen deficiency. However, these parameters have not been properly studied in a well-defined group of women with hypopituitarism. These baseline studies are needed prior to undertaking a study on treating women with hypopituitarism with a testosterone preparation.

Prior to investigating testosterone replacement in a large study of women with hypopituitarism, we must first determine in this pilot study the amount and interval of testosterone administration.

Currently, the only FDA-approved drug for testosterone in women is Estratest, which contains methyl testosterone, a compound that when given orally is associated with liver toxicity in animals and humans. Until recently, most hypogonadal men received biweekly intramuscular injections of testosterone. This regimen gives variable serum testosterone levels depending on the time of the blood sampling compared to the time of injection. Many male hypogonadal patients now receive their testosterone replacement via either transdermal testosterone gel or patch, with much more uniform serum testosterone levels. We have chosen transdermal testosterone gel for use in this study for several reasons:

1. Recent studies have shown that stable, reproducible levels of serum testosterone can be obtained irrespective of application site in hypogonadal men. No skin irritation (which can be problematic with the testosterone patch) was observed.
2. Graded Double-blinded dosing can easily be implemented.

Thus, we will use transdermal testosterone gel as it provides predictable and physiologic levels of testosterone.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18-55
* Hypopituitarism with documented central adrenal and gonadal deficiencies. Serum testosterone level of < 20 ng/dl or free testosterone <1.5 pg/ml on conjugated equine estrogen replacement
* No other significant medical condition
* Weight between 80 and 150% of ideal body weight
* Able to provide informed consent
* All races and ethnicities
* All patients regardless of marital status and relationship status

Exclusion Criteria:

* Physical disabilities that would prevent them from participating in the study
* Current use of testosterone or other androgenic steroids. Patients who are taking testosterone, DHEA or other androgen precursors will discontinue these medications/supplements three months prior to the study.
* Significant cardiopulmonary disease, renal disease (creatinine > 1.5 mg/dL), diabetes mellitus, uncontrolled hypertension, malignancy (other than basal cell skin carcinoma) or major psychiatric disease. Patients with depression or anxiety on a stable dose of medication will be allowed to enroll.
* Current abuse of illicit drugs or heavy ethanol use
* History of breast or uterine cancer
* Those with significant liver function abnormalities defined as SGOT, SGPT or alkaline phosphatase value of greater than one and one-half times the upper limit of normal in our Clinical Pathology Laboratory or serum bilirubin levels of greater than 2 mg/dl will be excluded.
* Those with history of hyperandrogenic disorders such as hirsutism and polycystic ovary disease will be excluded. These conditions are rare in women with hypopituitarism. Testosterone administration to these patients may exacerbate the underlying disorder.
* Women who are pregnant, seeking to become pregnant in the next 6 months, or breast feeding
* Those who have previously experienced intolerance to other transdermal systems
* Drugs known to alter testosterone production such as Megace or ketoconazole
* Patients with untreated hyperprolactinemia or active Cushing's disease. Patients with treated prolactinoma or Cushing's disease will be allowed to participate in the study.
* Hematocrit > 50%
* Male sex
* Not willing to answer all questions on surveys

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2002-08; Primary Completion 2002-08 (Actual); Study Completion 2002-08 (Actual)

PRIMARY OUTCOMES:
The purpose of this study is to determine the pharmacokinetics of testosterone gel 2 mg/d administered for a week to women with hypopituitarism and determine if this leads to testosterone replacement in a physiologic range. | 6 weeks

SECONDARY OUTCOMES:
An additional objective is to determine the baseline laboratory abnormalities and physical, cognitive, emotional and sexual symptomatology of these women with hypopituitarism. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ted C Friedman, M.D., Ph.D., Principal Investigator — Charles Drew University of Medicine and Science
Locations (1):
- Charles R. Drew University, Los Angeles, California, United States

REFERENCES:
- See also: Clinical Trial Research site — http://www.centerwatch.com